CLINICAL TRIAL: NCT01263548
Title: To Evaluate the Safety and Metabolic Profile of Vyvanse for the Treatment of ADHD in Euthymic Adults With Bipolar I/II Disorder
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Other Study IDs: Vyvanse-BD
Record Dates: First submitted 2010-12-14; First posted 2010-12-20 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Attention Deficit/Hyperactivity Disorder; Bipolar Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Bipolar Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Vyvanse: This is an open-label study which means that all study participants will be taking active study medication, Vyvanse.
  Interventions: Drug: lisdexamfetamine dimesylate

INTERVENTIONS:
Drug: lisdexamfetamine dimesylate — Dosage form: Capsules; Dosage strength: 30-70mg/day, flexible dosing; Duration: 4 weeks
  Other Names: Vyvanse

SUMMARY:
ADHD in the adult population is associated with several measures of harmful dysfunction. For example, adult ADHD is associated with high rates of separation/divorce and never-married status, lower educational attainment and occupational achievement, absenteeism, presenteeism, and job termination, as well as decreased social function. Individuals with adult ADHD are more likely than controls to have a comorbid diagnosis of bipolar disorder, alcohol and substance abuse, as well as antisocial personality disorder.

Psychostimulants are the most frequently employed medications in the treatment of adult ADHD. Several psychostimulants are Health Canada and US FDA-approved for the treatment of ADHD symptoms in adulthood.

Hitherto, no trial has evaluated the safety and efficacy of a psychostimulant in the treatment of ADHD symptomatology in adult individuals with bipolar disorder.

Vyvanse is the first prodrug stimulant indicated for the treatment of adult (and pediatric) ADHD. Vyvanse is a therapeutically inactive molecule (i.e. prodrug). After oral ingestion, lisdexamfetamine is converted to l-lysine, a naturally occurring essential amino acid, and active d-amphetamine, which is responsible for the drug's activity. Vyvanse provides a longer duration of effect consistent throughout the day with reduced potential for risk of abuse. Vyvanse is generally well tolerated with an adverse event profile similar to other psychostimulant medications. Available evidence indicates that in most treated subjects, Vyvanse is weight-neutral and/or is associated with weight loss. Moreover, in some individuals, it is associated with improvement in both glucose and lipid homeostasis.

The evaluation of safety/tolerability profiles as well as the effectiveness of lisdexamfetamine in a "real-world" population has significant translational value.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient status
* Male or female subjects between the ages of 18 to 55 years, inclusive
* Primary diagnosis of Bipolar Disorder and ADHD according to criteria in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) using the Mini International Neuropsychiatric Interview.
* Agree to use reliable method of birth control
* YMRS score </= 12
* CGI-BP < 6
* Able and willing to provide a written informed consent

Exclusion Criteria:

* Current Axis I primary psychiatric diagnosis other than Bipolar Disorder and ADHD
* Current Axis II psychiatric disorder of primary clinical focus
* Active alcohol as well as illicit or other substance abuse during the past 3 months
* Current clinically unstable medical condition.
* Inability to understand and engage in the process of informed consent.
* Inability to cooperate with study procedures.
* Presence of known allergies or hypersensitivity to lisdexamfetamine
* History of destabilization when exposed to psychostimulant medication
* Current high risk of suicide
* Current treatment with corticosteroids
* Electroconvulsive therapy in the last 1 year
* Current participation in a separate clinical research study involving an investigational drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals who have a diagnosis of Bipolar Disorder and ADHD.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Metabolic parameters | Screening (Week -1) to Endpoint (Week 4); Completed weekly on all 6 visits
  Weight; BMI; Waist circumference

SECONDARY OUTCOMES:
ADHD-RS | Baseline (Week 0) to Endpoint (Week 4); completed weekly on 5 visits
  Measure of ADHD symptoms
CAARS | Baseline (Week 0) to Endpoint (Week 4); completed weekly on 5 visits
  Measure of ADHD symptoms
CGI-BP | Baseline (Week 0) to Endpoint (Week 4); Completed weekly on all 6 visits
Q-LES-Q | Baseline (Week 0) and Endpoint (Week 4); Completed on 2 visits
  Quality of Life
AAQoL | Baseline (Week 0), Week 2, Endpoint (Week 4); Completed on 3 visits
  Quality of Life
Metabolic Peptidergic systems | Baseline (Week 0) and Endpoint (Week 4); Completed on 2 visits
  Insulin; Resistin; Ghrelin; Leptin; Adiponectin

CONTACTS AND LOCATIONS:
Locations (1):
- Mood Disorders Psychopharmacology Unit, Toronto, Ontario, Canada